CLINICAL TRIAL: NCT02570984
Title: Controlling and Preventing Asthma Progression and Severity in Kids
Brief Title: Preventing Asthma in High Risk Kids
Acronym: PARK
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Wanda Phipatanakul, Professor of Pediatrics, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB-P00019640; U01AI179563 (NIH)
Record Dates: First submitted 2015-07-28; First posted 2015-10-08 (Estimated); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): omalizumab 0.016 mg/kg/IU total IgE
  Interventions: Drug: Omalizumab
- Placebo (Placebo Comparator): looks like active drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omalizumab — anti-ige injection
  Other Names: Xolair
  Arms: Active
Drug: Placebo — placebo comparator arm, injection similar to active
  Other Names: placebo arm
  Arms: Placebo

SUMMARY:
This trial is a randomized, double-blind, placebo controlled trial designed to test whether two years treatment of preschool children aged 2-3 years of age at high risk for asthma with omalizumab (anti-IgE) for two years will prevent the progression to childhood asthma, as reflected by a reduction in the prevalence of active asthma in the Final 12 months during 2 year observation period off study drug.

DETAILED DESCRIPTION:
Prevention/ Disease modification of asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Parent/guardian must be able to understand and provide signed and dated written informed consent; he/she must also be able to communicate with study staff.
2. 24-47 months of age at randomization
3. 2-4 wheezing episodes in the past year
4. positive allergy to aeroallergen
5. first degree relative with history or current diagnosis of asthma or allergy
6. If is participating in a food immunotherapy treatment that is not part of a clinical trial, has been on an established maintenance regimen implemented continuously for a minimum of 2 months.

Exclusion Criteria:

1. >4 episodes of wheezing in the past year
2. Use of Step 5 or Step 6 therapy (ICS plus LABA ) at the time of enrollment (Visit 0).
3. Need for systemic corticosteroids or a hospitalization for respiratory symptoms within four weeks prior to screening.
4. Three or more courses of systemic corticosteroids for wheezing illnesses in the last year
5. More than four days of symptoms of wheezing, or tightness in the chest or cough in the past two weeks causing at least minimal limitation of activity
6. More than four days of albuterol treatment (for symptoms) in the past two weeks
7. More than one night of symptoms of wheezing, or tightness in the chest or cough causing sleep disruption in the past two weeks
8. More than one night of albuterol treatment (for symptoms) in the past two weeks
9. Prematurity (<34 weeks gestation)
10. Need for oxygen for more than 5 days in the neonatal period
11. History of intubation or mechanical ventilation for respiratory illness
12. Other significant medical conditions, including: major congenital anomalies, cystic fibrosis, chronic pulmonary diseases, bronchopulmonary dysplasia, thoracic surgery, history of tuberculosis, immunodeficiency (primary or secondary), seizure disorders
13. Expecting to relocate within 4 years of study initiation to a place which would make in-person clinical visits impossible
14. Deemed unable to adhere to study activities
15. Prior aeroallergen immunotherapy or use of biologics including anti-IgE
16. Prior IVIG or systemic immunosuppressant other than corticosteroids
17. History of hypoxic seizures during a wheezing episode
18. Total IgE outside of the omalizumab dosing range.
19. Enrolled in any clinical medication trial within the past 30 days.
20. With platelet counts < 150 x 109/L at the Screening Visit (V0)
21. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or may impact the quality or interpretation of the data obtained from the study.
22. History of severe anaphylactic/anaphylactoid reactions from any cause

Ages: 24 Months to 47 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2018-11-27 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
active asthma diagnosis | Final 12 months during 2 year observation period off study drug
  questionnaire
asthma severity | Final 12 months during 2 year observation period off study drug
  questionnaire

SECONDARY OUTCOMES:
number of positive new allergic sensitization | Final 12 months during 2 year observation period off study drug
  skin prick test
decrease in number of wheezing episodes | Final 12 months during 2 year observation period off study drug
  questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Wanda Phipatanakul, MD, MS, Principal Investigator — Boston Children's Hospital
Locations (13):
- United States (13):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Rady Children's Hospital - San Diego, San Diego, California
  - Childrens Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Hospital, Hartford, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Indiana University/Riley Children's Hospital, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Texas Children's Hospital/Baylor College of Medicine, Houston, Texas
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Derived] Phipatanakul W, Mauger DT, Guilbert TW, Bacharier LB, Durrani S, Jackson DJ, Martinez FD, Fitzpatrick AM, Cunningham A, Kunselman S, Wheatley LM, Bauer C, Davis CM, Geng B, Kloepfer KM, Lapin C, Liu AH, Pongracic JA, Teach SJ, Chmiel J, Gaffin JM, Greenhawt M, Gupta MR, Lai PS, Lemanske RF, Morgan WJ, Sheehan WJ, Stokes J, Thorne PS, Oettgen HC, Israel E; PARK Study Team. Preventing asthma in high risk kids (PARK) with omalizumab: Design, rationale, methods, lessons learned and adaptation. Contemp Clin Trials. 2021 Jan;100:106228. doi: 10.1016/j.cct.2020.106228. Epub 2020 Nov 24. PMID 33242697
- [Derived] Martinez FD. Childhood Asthma Inception and Progression: Role of Microbial Exposures, Susceptibility to Viruses and Early Allergic Sensitization. Immunol Allergy Clin North Am. 2019 May;39(2):141-150. doi: 10.1016/j.iac.2018.12.001. PMID 30954166